CLINICAL TRIAL: NCT02338986
Title: Collection of Plasma From Subjects That Recovered From or Were Vaccinated To Emerging Infectious Diseases
Brief Title: Collection of Plasma From People Who Recovered From or Were Vaccinated to Emerging Infectious Diseases
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150056; 15-I-0056; NCT02406378 (obsolete NCT alias)
Record Dates: First submitted 2015-01-14; First posted 2015-01-15 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Communicable Diseases; Communicable Diseases, Emerging; Emerging Infectious Diseases; Infection
Keywords: High Titer Antibodies; Convalescent Volunteers; Apheresis; Males; Quantitative IgG; Natural History
MeSH Terms: conditions — Communicable Diseases; Communicable Diseases, Emerging; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Collection of Plasma From Subjects That Recovered From or Were Vaccinated To Emerging Infectious Diseases
  Interventions: Drug: Plasma

INTERVENTIONS:
Drug: Plasma — Plasma

SUMMARY:
Background:

- There are more emerging infectious diseases recently. Some could affect many people. Some like Severe Acute Respiratory Syndrome (SARS) or Middle East Respiratory Syndrome (MERS) are caused by new germs. Sometimes known germs suddenly infect new and large areas, like Ebola. Many of these diseases don t have good treatments available. Researchers may be able to develop a treatment by using antibodies against these infections.

Objective:

- To collect antibodies from people with high levels of antibodies to the diseases being studied.

Eligibility:

- Ages 18-70 years old who weigh at least 110 pounds. They may have been infected with or vaccinated for one of the new infections researchers are studying.

Design:

* Participants will be screened with medical history and blood tests. Researchers will determine if the participant can have apheresis.
* Participants will have apheresis. First, they will be interviewed. Then, a needle will be placed in a vein. Blood will be drawn, and a machine will separate the blood cells from the antibodies and protein. The blood cells will then be returned to the participant through another vein. It takes about 60 minutes for the actual collection.
* Participants will be asked to have the procedure at least 3 times. They can participate in up to 20 sessions total as part of this study. There must be at least 7 days between sessions.

DETAILED DESCRIPTION:
The administration of convalescent plasma is often used for treatment of emerging infectious diseases. This natural history protocol will collect plasma from subjects that were vaccinated to or recovered from an emerging infectious disease of interest, in a manner that the plasma can be given to other subjects as a therapeutic. Any administration of plasma to subjects will be under a separate protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Provide written informed consent before initiation of any study procedures
  2. Age >=8 years old, and <=70 years old
  3. History of a known infection or vaccination towards emerging infectious diseases of interest:
* For convalescent subjects, the following criteria must be met:

  * At least 28 days since the subject was symptomatic from the infection
  * Afebrile (subjective history acceptable) for at least 28 days
  * Enrollment must occur within 24 months of illness.
* For vaccinated subjects, the following criteria must be met:

  * Subjects must be at least 14 days after vaccination
  * If vaccinated on a blinded study, the study must be unblinded and the subject received active product.
  * Enrollment must occur within 24 months of the last vaccination.
  * (The above represent the minimum criteria - more restrictive criteria may be listed under disease specific criteria noted in Appendix A)

    4) Weight >=110 pounds (50 kg)

    5) Adequate peripheral venous access for plasma donation (as judged by the examiner)

    6) Willingness to have samples stored

EXCLUSION CRITERIA:

1. Any sign of active infection (as judged by the investigator), including but not limited

   to:
   * Subjective or documented fever (>38 (Infinite)C)
   * Cough
   * Shortness of breath
   * Diarrhea
2. Pregnancy
3. Meets current blood establishment plasma donation exclusion criteria. A protocol amendment will not be needed to reflect updated/current blood donation exclusion criteria.
4. Subjects that have participated in previous plasma collection or other cell component collection procedures within the last 3 months may have restrictions to participation based on the site plasma collection standard operating procedure (SOP). In this scenario, discussion should occur with the blood establishment to ensure eligibility to donate plasma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women who have high titer antibodies for a given emerging infectious disease.@@@
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Number of units of plasma collected | 5 years after enrollment
  The number of units of human plasma collected from volunteers with high titer antibodies for a given emerging infectious disease, that is potentially suitable for infusion into humans as part of a separate treatment study.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Davey, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Soo YO, Cheng Y, Wong R, Hui DS, Lee CK, Tsang KK, Ng MH, Chan P, Cheng G, Sung JJ. Retrospective comparison of convalescent plasma with continuing high-dose methylprednisolone treatment in SARS patients. Clin Microbiol Infect. 2004 Jul;10(7):676-8. doi: 10.1111/j.1469-0691.2004.00956.x. PMID 15214887
- [Background] Mupapa K, Massamba M, Kibadi K, Kuvula K, Bwaka A, Kipasa M, Colebunders R, Muyembe-Tamfum JJ. Treatment of Ebola hemorrhagic fever with blood transfusions from convalescent patients. International Scientific and Technical Committee. J Infect Dis. 1999 Feb;179 Suppl 1:S18-23. doi: 10.1086/514298. PMID 9988160
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-I-0056.html